CLINICAL TRIAL: NCT05928299
Title: Proteomic and Metabolomic Features Testing for Immunotherapy Response in Non-Small Cell Lung Cancer
Brief Title: Integrative Multi-Omics Testing for Immunotherapy Response in Non-Small Cell Lung Cancer
Acronym: IMOTION
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2023-128
Record Dates: First submitted 2023-05-08; First posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Lung Cancer
Keywords: Non-Small Cell Lung Cancer; Immunotherapy; Blood Proteomic; Blood Metabolomic; Urine Proteomic; Urine Metabolomic; Monitoring of Immunotherapy Response; Multi-omics
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Durable Clinical Benefit: PFS≥ 6 months
- Non-durable Clinical Benefit: PFS< 6 months

SUMMARY:
The objective of this study is to use blood and urine proteomic and metabolomic features to monitor lung cancer immunotherapy response.

DETAILED DESCRIPTION:
Observational, ambispective single-center cohort study, including 400 patients with locally advanced unresectable or metastatic NSCLC who received or are receiving immunotherapy in routinely clinical practice.

For the part of retrospective study，the investigators intend to include 200 patients who received immunotherapy at Nanfang Hospital from January 1, 2020 to March 1, 2023.

For the part of prospective study，the investigators intend to include 200 patients who will receive immunotherapy at Nanfang Hospital from March 1, 2023 to December 31, 2025.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are 18 years or older at the time of signing the informed consent form;
2. Patients with histologically or cytologically confirmed non-small cell lung cancer that is metastatic or locally advanced unresectable, not eligible for local curative treatment (Stage IIIB or IV according to AJCC);
3. Patients without contraindications for immunotherapy according to CSCO guidelines for Non-Small Cell Lung Cancer (NSCLC) version 2022（No EGFR mutations, ALK or ROS1 rearrangement);
4. Patients with at least one measurable lesion according to the Response Evaluation Criteria in Solid Tumors [RECIST], version 1.1;
5. Patients who have not received systemic treatment in the past, or who have previously received (neo) adjuvant treatment/radical treatment programs and have relapsed for more than 6 months;
6. Patients who signed the informed consent and are willing to participate in the study.

Exclusion Criteria:

1. Patients with the history of autoimmune disease or immunodeficiency disease;
2. Any severe, uncontrolled diseases, including: (1) Active or uncontrolled heart diseases, (2) Renal failure requires hemodialysis or peritoneal dialysis; (3) Liver diseases such as liver cirrhosis, decompensated liver disease, chronic active hepatitis;
3. Any severe, uncontrolled urological diseases, or urine total protein >1.0g/day.
4. Any severe, uncontrolled metabolic diseases, including uncontrolled diabetes mellitus (fasting blood glucose (FBG)>10mmol/L);

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced NSCLC eligible for treatment of immunotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The expression of blood and urine proteomic markers at baseline | Baseline
  Blood and urine proteins detected by nanoparticle-based mass spectrometry at baseline. Proteins identified by the proteomic assay will include but will not be limited to KRAS, CCL5, CXCL12 and ANGPTL6.
The levels of blood and urine metabolites at baseline | Baseline
  Blood and urine metabolites detected by mass spectrometry and nuclear magnetic resonance at baseline. Metabolites identified by the metabolic assay will include but will not be limited to methionine, lactic acid and LDL-C
The expression of blood and urine proteomic markers during immunotherapy | 3 years
  Blood and urine proteins detected by nanoparticle-based mass spectrometry during immunotherapy. Proteins identified by the proteomic assay will include but will not be limited to KRAS, CCL5, CXCL12 and ANGPTL6.
The levels of blood and urine metabolites during immunotherapy | 3 years
  Blood and urine metabolites detected by mass spectrometry and nuclear magnetic resonance during immunotherapy. Metabolites identified by the metabolic assay will include but will not be limited to methionine, lactic acid and LDL-C
The expression of blood and urine proteomic markers at progression | 3 years
  Blood and urine proteins detected by nanoparticle-based mass spectrometry at progression. Proteins identified by the proteomic assay will include but will not be limited to KRAS, CCL5, CXCL12 and ANGPTL6.
The levels of blood and urine metabolites at progression | 3 years
  Blood and urine metabolites detected by mass spectrometry and nuclear magnetic resonance at progression. Metabolites identified by the metabolic assay will include but will not be limited to methionine, lactic acid and LDL-C

SECONDARY OUTCOMES:
Immune-related adverse events (irAEs) | 3 years
  Immune-related adverse events (irAEs), as assessed by Common Terminology Criteria for Adverse Events (CTCAE - Version 5.0)

CONTACTS AND LOCATIONS:
Locations (1):
- Nanfang hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No